CLINICAL TRIAL: NCT00947453
Title: The Effect of Montelukast Therapy on mRNA Profile of Matrix Metalloproteinases and Their Inhibitors in the Sputum of Patients With Asthma
Brief Title: Sputum Matrix Metalloproteinases (MMP) mRNA and Montelukast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Dr Andrew M Wilson, University of East Anglia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009RESP01; EudraCT Number: 2008-008364-27
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: asthma; montelukast
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- montelukast group (Experimental): Identified patients with asthma to recieve Montelukast 10 mg (Merck Sharp & Dohme Ltd, Herts, UK) at 0800 am once daily for 8 weeks.
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: montelukast — montelukast 10 mg once daily for 8 weeks

SUMMARY:
Matrix metalloproteinases (MMPs) are a group of 24 zinc containing enzymes in man. These enzymes were originally described as cleaving extracellular matrix (ECM) substrates with a predominant role in ECM homeostasis, but it is now clear that they have much wider functionality. An imbalance between MMP activity and that of their inhibitors (tissue inhibitors of metalloproteinases, TIMPs) is considered to play a critical role in the synthesis or degradation of the extracellular matrix of the airway architecture which results in fixed airflow obstruction in both asthma and chronic obstructive pulmonary disease (COPD). Using quantitative real time polymerase chain reaction (RT-PCR) the investigators have identified a difference between the level of steady state mRNA for MMP-9, MMP-14 and MMP-2 in 2 patients with asthma compared to 4 healthy controls using our method. However the investigators require further refinement of the process in order to optimise RNA quality and to evaluate the effect of montelukast across the entire family of MMPs and their inhibitors (TIMPs).

DETAILED DESCRIPTION:
The following measurements will be performed at screening:

* Informed consent
* Clinical examination
* Spirometry
* Induced sputum

The following will be performed after 8 weeks of study medication:

* Clinical examination
* Spirometry
* Induced sputum
* Diary Card

Spirometry:

This will be performed with a Microlab spirometer (Micro Medical Ltd, Rochester, Kent, UK). The procedure will be according to American Thoracic Society specifications(13).

Diary Card Data:

Patients will record their symptoms on a daily basis in the morning according to "cough", "breathlessness" and "wheeze" on a 4 point scale with 0=no symptoms and 3=maximal symptoms. A total symptom score will be calculated out of 12. Patients will also measure their peak expiratory flow on a daily basis in the morning and record the highest of three measurements. They will record that they have taken their study medication.

Sputum Induction & Examination:

Sputum will be obtained with hypertonic saline by the method described by Pizzichini et al(14) inhaling increasing concentrations of saline (3, 4 and 5%) each for 7 minutes, through a mouthpiece. After each period of inhalation, FEV1 will be measured for safety. Subjects will be asked to cough sputum into a sterile container. Total cell count of leukocytes will be obtained in a modified Neubauer haemocytometer. The cell viability will be determined by the trypan blue exclusion method. Four hundred non squamous cells will be counted in Wright-stained slides and the results will be expressed as a percentage and absolute number of the total non squamous count. Measurement of MMP-9, 12 TIMP-1 and TGFb will be performed in sputum supernatant.

Profile of mRNA of MMP and TIMPs:

Total RNA will be extracted from the cellular content of the induced sputum plug using a combination of Trizol extraction and Qiagen RNeasy spin columns in a similar way to previously described12. Quantitative RT-PCR, using previously developed primers and probes, will be used to determine the relative quantities of mRNA of MMPs and TIMPs as described12. We remain the only centre in the world to routinely profile the entire MMP and TIMP gene family in human samples. This gives an all encompassing view of the involvement of these enzymes and inhibitors in the disease process and also sheds light on potential new biomarkers. The possibility of expanding the gene profiling without the need for additional sputum collection also adds value to the research. This might include other proteinase families with roles in ECM breakdown or in inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 60 years.
* Diagnosed with asthma, defined as episodic chest tightness, wheezing and dyspnoea, cough.
* Non-Smoker or Ex-Smoker for at least 10 years and a smoking history of less than 5 pack years.
* History of asthma symptoms for more than 10years.
* Receiving as required short acting bronchodilators.
* Post bronchodilator FEV1 50 to 100 % predicted
* Evidence of airway calibre reversibility within the previous 12 months: reversibility to salbutamol of 12% following 400mcg inhaled salbutamol, histamine PC20 < 8mg/ml, diurnal variation in peak expiratory flow of 20%.
* Able to produce sputum after induction with saline.

Exclusion criteria:

* Cardiac or pulmonary disease other than asthma.
* Respiratory infection defined as fever, nasal/sinus congestion, fatigue, cough, antibiotic use or yellow/green sputum within 4 weeks prior to study.
* Receiving inhaled or oral corticosteroid therapy, long acting Beta2 agonist therapy or leukotriene modifying therapy for the previous 1 month.
* Severe or uncontrolled co-morbid disease.
* Pregnancy or breastfeeding.
* Unable to give written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the MMP and TIMP mRNA profile relative to a housekeeping gene | 8 weeks

SECONDARY OUTCOMES:
The difference between treatment with montelukast for 8 weeks and placebo for mRNA for MMP and TIMP | 8 weeks
The difference between treatment with montelukast for 8 weeks and placebo for Spirometry - FEV1, FVC, FEV1/FVC ratio | 8 weeks
The difference between treatment with montelukast for 8 weeks and placebo for Induced sputum differential cell count | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, MRCP (UK), Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Cauwe B, Van den Steen PE, Opdenakker G. The biochemical, biological, and pathological kaleidoscope of cell surface substrates processed by matrix metalloproteinases. Crit Rev Biochem Mol Biol. 2007 May-Jun;42(3):113-85. doi: 10.1080/10409230701340019. PMID 17562450
- [Background] Suzuki R, Miyazaki Y, Takagi K, Torii K, Taniguchi H. Matrix metalloproteinases in the pathogenesis of asthma and COPD: implications for therapy. Treat Respir Med. 2004;3(1):17-27. doi: 10.2165/00151829-200403010-00003. PMID 15174890
- [Background] Atkinson JJ, Senior RM. Matrix metalloproteinase-9 in lung remodeling. Am J Respir Cell Mol Biol. 2003 Jan;28(1):12-24. doi: 10.1165/rcmb.2002-0166TR. PMID 12495928
- [Background] Kelly EA, Busse WW, Jarjour NN. Increased matrix metalloproteinase-9 in the airway after allergen challenge. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1157-61. doi: 10.1164/ajrccm.162.3.9908016. PMID 10988146
- [Background] Boulay ME, Prince P, Deschesnes F, Chakir J, Boulet LP. Metalloproteinase-9 in induced sputum correlates with the severity of the late allergen-induced asthmatic response. Respiration. 2004 May-Jun;71(3):216-24. doi: 10.1159/000077418. PMID 15133340
- [Background] Beeh KM, Beier J, Kornmann O, Buhl R. Sputum matrix metalloproteinase-9, tissue inhibitor of metalloprotinease-1, and their molar ratio in patients with chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis and healthy subjects. Respir Med. 2003 Jun;97(6):634-9. doi: 10.1053/rmed.2003.1493. PMID 12814147
- [Background] Vignola AM, Riccobono L, Mirabella A, Profita M, Chanez P, Bellia V, Mautino G, D'accardi P, Bousquet J, Bonsignore G. Sputum metalloproteinase-9/tissue inhibitor of metalloproteinase-1 ratio correlates with airflow obstruction in asthma and chronic bronchitis. Am J Respir Crit Care Med. 1998 Dec;158(6):1945-50. doi: 10.1164/ajrccm.158.6.9803014. PMID 9847290
- [Background] Barnes PJ, Hansel TT. Prospects for new drugs for chronic obstructive pulmonary disease. Lancet. 2004 Sep 11-17;364(9438):985-96. doi: 10.1016/S0140-6736(04)17025-6. PMID 15364192
- [Background] Langlois A, Ferland C, Tremblay GM, Laviolette M. Montelukast regulates eosinophil protease activity through a leukotriene-independent mechanism. J Allergy Clin Immunol. 2006 Jul;118(1):113-9. doi: 10.1016/j.jaci.2006.03.010. Epub 2006 May 19. PMID 16815146
- [Background] Vignola AM, Riccobono L, Profita M, Foresi A, Di Giorgi R, Guerrera D, Gjomarkaj M, Di Blasi P, Paggiaro PL. Effects of low doses of inhaled fluticasone propionate on inflammation and remodelling in persistent-mild asthma. Allergy. 2005 Dec;60(12):1511-7. doi: 10.1111/j.1398-9995.2005.00827.x. PMID 16266383
- [Background] Chuang SS, Hung CH, Hua YM, Tien CH, Yang KD, Jong YJ, Hsu SH, Lin CS. Suppression of plasma matrix metalloproteinase-9 following montelukast treatment in childhood asthma. Pediatr Int. 2007 Dec;49(6):918-22. doi: 10.1111/j.1442-200X.2007.02497.x. PMID 18045297
- [Background] Kevorkian L, Young DA, Darrah C, Donell ST, Shepstone L, Porter S, Brockbank SM, Edwards DR, Parker AE, Clark IM. Expression profiling of metalloproteinases and their inhibitors in cartilage. Arthritis Rheum. 2004 Jan;50(1):131-41. doi: 10.1002/art.11433. PMID 14730609
- [Background] Standardization of spirometry--1987 update. Statement of the American Thoracic Society. Am Rev Respir Dis. 1987 Nov;136(5):1285-98. doi: 10.1164/ajrccm/136.5.1285. No abstract available. PMID 3674589
- [Background] Pizzichini E, Pizzichini MM, Efthimiadis A, Evans S, Morris MM, Squillace D, Gleich GJ, Dolovich J, Hargreave FE. Indices of airway inflammation in induced sputum: reproducibility and validity of cell and fluid-phase measurements. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):308-17. doi: 10.1164/ajrccm.154.2.8756799.